CLINICAL TRIAL: NCT03291483
Title: The Effects of Whole Body Vibration With Plyometric Training on Physical Performance in Basketball Players
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Günseli Usgu, Asistant professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO 15/427
Record Dates: First submitted 2017-09-01; First posted 2017-09-25 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Muscle Strength; Postural Balance; Range of Motion, Articular; Walking Speed, Mesh id D000072797
Keywords: Whole body vibration; mesh id D000072797; Plyometric exercise; Muscle strength; Physical fitness; Balance
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration group (Experimental): basketball players had done exercises on whole body vibration platform.
  Interventions: Other: whole body vibration; Other: plyometric training
- plyometric training (Sham Comparator): Basketball players had done same plyometric exercises
  Interventions: Other: plyometric training

INTERVENTIONS:
Other: whole body vibration — whole body vibration is a mechanical stimulus characterized by oscillatory movements.Whole body vibration's potential beneficial effects occurs by transmission of mechanical and sinusoidal vibrations to the whole body through the feet.
  Arms: whole body vibration group
Other: plyometric training — Plyometric exercises refers to performance of stretch-shortening cycle (SSC) movements that involve a high-intensity eccentric contraction immediately after a rapid and powerful concentric contraction.

SUMMARY:
Purpose: The purpose of this study was to determine whether whole body vibration with plyometric training has effect on physical performance parameters and balance also this study searched for if vibration support additional benefits to normal plyometric training. Methods: 24 elite basketball players divided into two group as 12 players with the mean age of 24 ± 6,96 years (Study Group) and 12 players with the mean age of 22,45 ± 5,22 years (Control Group). Plyometric training were applied to study group on whole body vibration platform for 6 weeks (2 days/week) with routine basketball training, in control group plyometric training were applied on whole body vibration platform with the similar period of time but platform had been closed. All the assessments (physical measurement, vertical and horizontal jump tests, one-repetition maximum (1-RM) half squat strength test, 20 m speed test, T agility test, sit and reach flexibility test, star excursion balance test) were applied before and after 6 weeks plyometric training for both groups.

ELIGIBILITY:
Inclusion Criteria:

* male basketball player
* professional basketball player
* age between 18-28

Exclusion Criteria:

* lower extremity injuries
* upper extremity injuries

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2016-08-13 (Actual)

PRIMARY OUTCOMES:
muscle strength | changes in muscle strength at 6 weeks later
  1 Repetition maximum half squat test
muscular power | changes in muscular power at 6 weeks later
  vertical jump test
flexibility | changes in flexibility at 6 weeks later
  sit and reach test
balance | changes in balance at 6 weeks later
  star excursion balance test

CONTACTS AND LOCATIONS:
Overall Officials: Günseli Usgu, asst. prof., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Preatoni E, Colombo A, Verga M, Galvani C, Faina M, Rodano R, Preatoni E, Cardinale M. The effects of whole-body vibration in isolation or combined with strength training in female athletes. J Strength Cond Res. 2012 Sep;26(9):2495-506. doi: 10.1519/JSC.0b013e31823f299d. PMID 22067255
- [Background] Kurt C, Pekunlu E. Acute effect of whole body vibration on isometric strength, squat jump, and flexibility in well-trained combat athletes. Biol Sport. 2015 Jun;32(2):115-22. doi: 10.5604/20831862.1134558. Epub 2015 Jan 14. PMID 26060334
- [Background] Colson SS, Pensini M, Espinosa J, Garrandes F, Legros P. Whole-body vibration training effects on the physical performance of basketball players. J Strength Cond Res. 2010 Apr;24(4):999-1006. doi: 10.1519/JSC.0b013e3181c7bf10. PMID 20300027
- [Background] Fagnani F, Giombini A, Di Cesare A, Pigozzi F, Di Salvo V. The effects of a whole-body vibration program on muscle performance and flexibility in female athletes. Am J Phys Med Rehabil. 2006 Dec;85(12):956-62. doi: 10.1097/01.phm.0000247652.94486.92. PMID 17117001
- [Background] Despina T, George D, George T, Sotiris P, Alessandra DC, George K, Maria R, Stavros K. Short-term effect of whole-body vibration training on balance, flexibility and lower limb explosive strength in elite rhythmic gymnasts. Hum Mov Sci. 2014 Feb;33:149-58. doi: 10.1016/j.humov.2013.07.023. Epub 2013 Sep 20. PMID 24055361
- [Background] Arazi, H., Asadi, A. (2011 ). The effect of aquatic and land plyometric training on strength, sprint, and balance in young basketball players. Journal of human sport & exercise, 6 (1 ), 101-111.
- [Background] Bullock N, Martin DT, Ross A, Rosemond CD, Jordan MJ, Marino FE. Acute effect of whole-body vibration on sprint and jumping performance in elite skeleton athletes. J Strength Cond Res. 2008 Jul;22(4):1371-4. doi: 10.1519/JSC.0b013e31816a44b5. PMID 18545165